CLINICAL TRIAL: NCT07319273
Title: Application of Child Life Services in Pediatric Skin Prick Test
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHFudanU1013
Record Dates: First submitted 2025-11-16; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Hypersensitivity; Pediatrics
Keywords: child life services; skin prick test; pain; anxiety; pediatric nursing
MeSH Terms: conditions — Hypersensitivity; Pain; Anxiety Disorders | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups (intervention or control) based on visit time, with each group receiving a single intervention throughout the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): Receive standard care during the skin prick test.
  Interventions: Behavioral: Standard Care (in control arm)
- Child life services (Experimental): Receive child life services during the skin prick test.
  Interventions: Behavioral: child life services

INTERVENTIONS:
Behavioral: Standard Care (in control arm) — Nurses introduce the environment, personnel, and procedure, review the child's medical and allergy history, and confirm informed consent. The SPT is then performed according to clinical standards. After the procedure, children remain under observation, during which nurses monitor for any discomfort and provide guidance to avoid scratching the test site. Finally, nurses measure and interpret the results and provide basic health education to the child and caregivers.
  Arms: Standard of care
Behavioral: child life services — Children in the intervention group receive standard care plus support from a Child Life Specialist (CLS) throughout the SPT procedure. The CLS provides age-appropriate preparation, distraction, and emotional support to both children and caregivers before, during, and after the procedure. The CLS also monitors the child's responses, helps manage any anxiety or resistance, supports caregivers emotionally, and explains test results and post-procedure care in an understandable manner.
  Arms: Child life services

SUMMARY:
The goal of this clinical trial is to determine whether child life services can enhance the experiences of children and caregivers during skin prick testing. The main questions it aims to answer are:

1. Can child life services alleviate children's pain and enhance procedural compliance?
2. Can child life services reduce caregivers' anxiety and improve their satisfaction? Researchers will compare children who receive child life services with those who receive standard care to determine whether the intervention can optimize procedural experience and overall satisfaction.

Participants will receive either child life services or standard care during the skin prick test.

DETAILED DESCRIPTION:
The skin prick test (SPT) is an essential diagnostic tool for IgE-mediated allergic diseases and a foundation for allergen immunotherapy. However, the multiple needle pricks involved often cause pain and anxiety in children, while caregivers frequently experience heightened stress. Child life services aim to help children feel safe and relaxed in medical settings, thereby reducing distress and improving cooperation. This study applied child life services during pediatric SPT to alleviate children's pain, boost procedural compliance, reduce procedural duration and interruptions, and enhance caregiver satisfaction while alleviating their anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Meet the indications for skin prick test (SPT)
* Aged 1-18 years
* Voluntarily agree to participate in the study and provide informed consent

Exclusion Criteria:

* Meet the contraindications for SPT
* Presence of psychiatric disorders or cognitive impairment
* Severe dysfunction of vital organs such as the heart, brain, or kidneys

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
the Face, Legs, Activity, Cry, Consolability (FLACC) scale score | Periprocedural
  Use the FLACC scale to assess pain, higher scores indicate greater pain (0 no pain, 1-3 mild pain, 4-6 moderate pain, 7-10 severe pain).
the Wong-Baker FACES score | Periprocedural
  Use the Wong-Baker FACES scale to assess pain, higher scores indicate greater pain (0 no pain, 1-3 mild pain, 4-6 moderate pain, 7-10 severe pain).
the Visual Analogue Scale (VAS) score | Periprocedural
  Use the Visual Analogue Scale (VAS) to assess pain, higher scores indicate greater pain (0 no pain, 1-3 mild pain, 4-6 moderate pain, 7-10 severe pain).
Child procedural compliance | Periprocedural
  During the skin-prick test, compliance was rated as:
  Full: complete cooperation with the nurse; Partial: test completed despite crying or resistance; None: test impossible owing to non-copliance Overall compliance rate = (full + partial) / total × 100%. A higher overall compliance rate indicates better overall compliance with the skin-prick test procedure.

SECONDARY OUTCOMES:
Procedure duration | Periprocedural
Number of interruptions | Periprocedural
Caregiver anxiety | within 10 minutes after skin-prick test
  Caregiver anxiety was assessed with the 10-item short-form State-Trait Anxiety Inventory (five state and five trait items); each item is scored 1-4, with higher total scores indicating greater anxiety (Cronbach's α = 0.918).
Caregiver satisfaction | within 10 minutes after skin-prick test
  satisfaction was rated by caregivers on a 5-point scale: 5 = very satisfied, 4 = satisfied, 3 = neutral, 2 = dissatisfied, 1 = very dissatisfied.

IPD SHARING:
Plan to Share IPD: No